CLINICAL TRIAL: NCT03454217
Title: Impact of Tramadol and Oxycodone on Sleep Apnea
Acronym: TROXAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program director of regional anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CER 2017-01976
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Oxycodone; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone (Active Comparator): Postoperative pain treatment with oxycodone
  Interventions: Drug: Oxycodone
- Tramadol (Active Comparator): Postoperative pain treatment with tramadol
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Oxycodone — Postoperative pain treatment with oxycodone
  Arms: Oxycodone
Drug: Tramadol — Postoperative pain treatment with tramadol
  Arms: Tramadol

SUMMARY:
Postoperative pain is usually treated with opioids. Among them, oxycodone is popular in the daily practice as it is administered orally and is easily titrated. However, side-effects include increase duration and frequency of apneic episodes. Some authors believe that tramadol has less impact on these apneic episodes during the first postoperative night, based on a trial that reported conclusive results only during the first 2 postoperative hours. The objective of this randomized controlled trial is to compare the effect of postoperative pain treatment of oxycodone with tramadol on apneic episodes during the first and third postoperative nights.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for orthopaedic surgery on the lower limb under a spinal anaesthesia
* physical status I-III

Exclusion Criteria:

* planned surgical duration more than 3 hours
* contraindication to spinal anaesthesia
* severe respiratory disease
* patient treated for sleep apnea syndrome
* allergy to tramadol or oxycodone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index while lying supine | Postoperative night 1
  Apnea hypopnea index while lying supine

SECONDARY OUTCOMES:
Apnea hypopnea index in another position than supine | Postoperative night 1
Mean pulse oxymetry | Postoperative night 1
Apnea hypopnea index while lying supine | Postoperative night 3
Apnea hypopnea index in another position than supine | Postoperative night 3
Mean pulse oxymetry | Postoperative night 3
Pains scores (numeric rating scale) | Postoperative day 0, 1, 2 and 3
Opioid (oxycodone or tramadol) consumption | Postoperative day 0, 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Albrecht E, Pereira P, Bayon V, Berger M, Wegrzyn J, Antoniadis A, Heinzer R. The Relationship Between Postoperative Opioid Analgesia and Sleep Apnea Severity in Patients Undergoing Hip Arthroplasty: A Randomized, Controlled, Triple-Blinded Trial. Nat Sci Sleep. 2022 Feb 25;14:303-310. doi: 10.2147/NSS.S348834. eCollection 2022. PMID 35241942